CLINICAL TRIAL: NCT03008746
Title: Pulmonary Microbiota in COPD Patients Colonized With P. Aeruginosa OprD Mutant Resistant to Imipenem
Brief Title: Pulmonary Microbiota in Patients With Chronic Obstructive Pulmonary Disease Colonized With P. Aeruginosa Resistant to Imipenem
Acronym: MiPAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PA16090*
Record Dates: First submitted 2016-12-27; First posted 2017-01-02 (Estimated); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Therapeutic Irrigation

ARMS (3):
- not Pseudomonas aeruginosa colonized (Experimental)
  Interventions: Other: water used for oral wash; Other: sputum; Other: oral wash
- Pseudomonas aeruginosa colonized (Experimental)
  Interventions: Other: water used for oral wash; Other: sputum; Other: oral wash
- Pseudomonas aeruginosa OprD mutant colonized (Experimental)
  Interventions: Other: water used for oral wash; Other: sputum; Other: oral wash

INTERVENTIONS:
Other: water used for oral wash
Other: sputum
Other: oral wash

SUMMARY:
Pseudomonas aeruginosa (PA ) is associated with chronic lung infections in patients with chronic obstructive pulmonary disease (COPD). Commensal flora (microbiota) in lung was recently described using high-throughput sequencing techniques (NGS). PA strains isolated during lung infection episodes of severe COPD patients often show resistance to antibiotics including imipenem that is mainly due to mutation in oprD. In collaboration with Harvard Medical School, the investigators have recently demonstrated that PA OprD mutant shows increased survival (fitness) and its virulence. This bacterium could be more likely to colonize. Colonization by PA OprD mutant could influence the pulmonary microbiota and may worsen disease evolution, particularly in terms of frequency of exacerbations. Our objective is to describe modification of pulmonary microbiota associated with PA colonization, including OprD PA mutant, in severe COPD patients. The investigators will correlate the microbiota modification to medical history. Stable severe COPD patients will be included. Three groups of patients will be sampled: 1) not PA colonized, 2) PA colonized and 3) PA OprD mutant colonized. Medical history will be recorded by the physician as usual and three samples will be performed: 1) sputum, 2) oral wash and 3) water used for oral wash. Regular bacterial culture will be performed and NGS will be performed also to characterize the microbiota.

DETAILED DESCRIPTION:
Patients: Severe COPD Patients (FEV/Forced vital capacity (FVC)<70% and in FEV<50% after bronchodilation) hospitalized in the pulmonology Department of the Reims Teaching Hospital. At the inclusion, patients should be stable. Inclusion of 20 patients needing 100 patients in total will require 24 months.The study of associated factors with colonization to PA and PA mutant OprD will be performed only for patients known to be not PA carrier. Microbiota characterization will be performed on all patients colonized with PA and on non PA colonized patients randomly selected. The analysis of of PA colonization influence on COPD evolution will be done 12 months after sampling for all patients included.

Evaluation criteria:

* Presence of P. aeruginosa resistance to imipenem (OprD mutation)
* Pulmonary microbiota: Determination of the bacterial load (total number of bacterium) and bacterial community diversity. Then, Opertional Taxonomic Unit (OTU) relative abundance will be analyzed at phylum, class, order and family level.
* Factors associated with colonization with PA and PA mutant OprD: antibiotics, corticosteroids, hospitalization during the year preceding the inclusion, severity of COPD, respiratory symptoms of cough and expectoration, exertional dyspnea assessed by questionnaire the modified Respiratory Medical Council (MMRC), co-morbidities.
* PA porting Influence and PA mutant OprD on changes to 12 months: the number of exacerbation, severity of exacerbations, number of hospitalization, quality of life assessed by the St George's respiratory questionnaire, death, evolution of ventilatory disorders obstructive.

Investigation:

* Proposal for participation to all eligible patients at a pulmonology consultation
* If participation of acceptance (signed informed consent form): 3 bacteriological samples: Sputum (usually done), oral wash with water before washing (made specifically for this study). No change in the patient's medical care (treatment, monitoring, etc ...). Clinical Data Collection: criteria for COPD, pulmonary function, dyspnea and sputum symptoms, assessed by the MMRC scale, quality of life assessed by St George's respiratory questionnaire, antibiotic therapy and hospitalization in the previous 12 months . Revaluation 12 months after sampling as part of the regular monitoring of patients (idem as previously). All the samples will be sent to the clinical laboratory of bacteriology (CHU Reims) as usually done for samples: separation of sample into 2 parts: 1 part stored at -80 ° C and 1 part commonly analyzed. Then, patients will be classified as PA or PA non colonized based on sputum analysis. Mutation in oprD will be characterized in a second step to classify patients as PA or PA OprD mutant carriers. Samples of all patients colonized with PA and on non PA colonized patients randomly selected which have been stored at -80°C will be sent to the "PEGASE" plateform of Institut Pasteur de Lille. Characterization of pulmonary microbiota will be performed by high-throughput sequencing on Illumina "MiSeq" allowing to reach 24 million reads in 2x300 bp paired-end.

ELIGIBILITY:
Inclusion Criteria:

* Severe COPD Patients (FEV/FVC<70% and in FEV<50% after bronchodilation) hospitalized in the pulmonology Department of the Reims Teaching Hospital.
* patients who agreed to participate in the study.
* patients affiliated to a social security scheme.

Exclusion Criteria:

* patients <18yo
* patients protected by the law.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2017-01-12 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2022-05-17 (Actual)

PRIMARY OUTCOMES:
Presence of P. aeruginosa resistance to imipenem (OprD mutation) | 12 months
Pulmonary microbiota | 12 months
questionnaire: the modified Respiratory Medical Council (MMRC) | 12 months
St George's respiratory questionnaire | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

REFERENCES:
- [Background] Audebert C, Even G, Cian A; Blastocystis Investigation Group; Loywick A, Merlin S, Viscogliosi E, Chabe M. Colonization with the enteric protozoa Blastocystis is associated with increased diversity of human gut bacterial microbiota. Sci Rep. 2016 May 5;6:25255. doi: 10.1038/srep25255. PMID 27147260
- [Background] Wang Z, Bafadhel M, Haldar K, Spivak A, Mayhew D, Miller BE, Tal-Singer R, Johnston SL, Ramsheh MY, Barer MR, Brightling CE, Brown JR. Lung microbiome dynamics in COPD exacerbations. Eur Respir J. 2016 Apr;47(4):1082-92. doi: 10.1183/13993003.01406-2015. Epub 2016 Feb 25. PMID 26917613